CLINICAL TRIAL: NCT01951599
Title: A Phase I, Open-label, Single-center, Sequential Design Study in Healthy Volunteers to Determine the Relative Bioavailability of Different Oral Formulations of AZD9291 and the Effect of Food
Brief Title: To Determine the Relative Bioavailability of Different Formulations of AZD9291 and the Effect of Food.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D5160C00005
Record Dates: First submitted 2013-09-24; First posted 2013-09-26 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteers
Keywords: Phase I, healthy, bioavailability, pharmacokinetics, safety, tolerability.
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- AZD9291 20mg (oral capsule fasted) (Experimental): Volunteers will receive AZD9291 20mg administered by mouth, as a capsule, in the fasted state.
  Interventions: Drug: AZD9291
- AZD9291 20mg (oral solution fasted) (Experimental): Volunteers will receive AZD9291 20mg administered by mouth, as a solution, in the fasted state.
  Interventions: Drug: AZD9291
- AZD9291 20mg (oral tablet fasted) (Experimental): Volunteers will receive AZD9291 20mg administered by mouth, as a tablet, in the fasted state.
  Interventions: Drug: AZD9291
- AZD9291 20mg (oral fasted) (Experimental): Volunteers will receive AZD9291 20mg administered by mouth, as a capsule or tablet in the fasted state.
  Interventions: Drug: AZD9291
- AZD9291 20mg (oral fed) (Experimental): Volunteers will receive AZD9291 20mg administered by mouth, as a capsule or tablet in the fed state.
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD9291 — Volunteers will receive a single 20-mg dose of AZD9291 as a capsule on day 1, in Part A, Period 1, in the fasted state. (Treatment A).
  Arms: AZD9291 20mg (oral capsule fasted)
Drug: AZD9291 — Volunteers will receive a single 20-mg dose of AZD9291 as a solution on day 1, in Part A, Period 2, in the fasted state. (Treatment B).
  Arms: AZD9291 20mg (oral solution fasted)
Drug: AZD9291 — Volunteers will receive a single 20-mg dose of AZD9291 as a tablet on day 1, in Part A, Period 3, in the fasted state. (Treatment C).
  Arms: AZD9291 20mg (oral tablet fasted)
Drug: AZD9291 — Volunteers will receive a single 20-mg dose of AZD9291 as a capsule or tablet on day 1, in Part B, Period 1, in the fasted state.
  Arms: AZD9291 20mg (oral fasted)
Drug: AZD9291 — Volunteers will receive a single 20-mg dose of AZD9291 as a capsule or tablet on day 1, in Part B, Period 2, in the fed state.
  Arms: AZD9291 20mg (oral fed)

SUMMARY:
To determine the relative bioavailability of different oral formulations of AZD9291 and the effect of food in healthy volunteers.

DETAILED DESCRIPTION:
A Phase I, Open-label, Single-center, Sequential Design Study in Healthy Volunteers to Determine the Relative Bioavailability of Different Oral Formulations of AZD9291 and the Effect of Food

ELIGIBILITY:
Inclusion Criteria:

1, Body mass index between 19 and 30 kg/m2 and weight at least 50 kg and no more than 100 kg. 2, Volunteers must be willing to use a condom, unless their partners are postmenopausal, surgically sterile, or using an effective hormonal method of contraception or intrauterine coil. 3. In addition, volunteers must agree to continue to take similar contraceptive precautions until 4 months after the last dose of AZD9291.

Exclusion Criteria:

1. Any clinically relevant abnormalities in physical examination, vital signs, hematology, clinical chemistry, urinalysis or ECG at baseline in the opinion of the Investigator.
2. Volunteers who have received live or live-attenuated vaccine in the 2 weeks prior to dosing.
3. History of severe allergy/hypersensitivity or or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to AZD9291, its excipients, or drugs with a similar chemical structure or class.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2014-06-04 (Actual); Study Completion 2014-06-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of AZD9291 and its metabolites, by assessment of maximum plasma concentration (Cmax) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post dose
  Curve taken during each of the 5 treatments

SECONDARY OUTCOMES:
Pharmacokinetics of AZD9291 and its metabolites by assessment of the area under the plasma concentration-time curve from zero to infinity (AUC) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post dose
  Curve taken during each of the 5 treatments
Pharmacokinetics of AZD9291 and its metabolites, by assessment of time to Cmax (tmax) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post dose
  Curve taken during each of the 5 treatments
Pharmacokinetics of AZD9291 and its metabolites, by assessment of Terminal rate constant (λz) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post dose
  Curve taken during each of the 5 treatments
Pharmacokinetics of AZD9291 and its metabolites, by assessment of Terminal half life (t1/2,λz) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post dose
  Curve taken during each of the 5 treatments
Pharmacokinetics of AZD9291 and its metabolites, by assessment of lag time before observation of quantifiable analyte concentrations in plasma (tlag) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post dose
  Curve taken during each of the 5 treatments
Pharmacokinetics of AZD9291 and its metabolites, by assessment of area under the plasma concentration-time curve from zero to time of last measurable concentration [AUC(0-t)] | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post dose
  Curve taken during each of the 5 treatments
Pharmacokinetics of AZD9291 and its metabolites, by assessment of area under the plasma concentration-time curve from zero to 72 hours [AUC(0-72)] | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post dose
  Curve taken during each of the 5 treatments
Pharmacokinetics of AZD9291 only, by assessment of apparent plasma clearance (CL/F). | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post dose
  Curve taken during each of the 5 treatments
Pharmacokinetics of AZD9291 only, apparent volume of distribution (Vz/F) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post dose
  Curve taken during each of the 5 treatments
Pharmacokinetics of AZD9291 parent to metabolite ratio (calculated for both Cmax and AUC). | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, 504 hours post dose
  Curve taken during each of the 5 treatments

OTHER OUTCOMES:
Safety variables (adverse events, physical exam, vital signs, ECG's, clinical laboratory safety tests, opthalmological examination) | Baseline (Day-1) to Day 28
  Assessments performed during each of the 5 treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Phil Leese, MD, Principal Investigator — Quintiles 6700 W 115th Street, Kansas, US
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- See also: D5160C00005revised_csp_2_signed_31March 16_REDACTED — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1901&filename=D5160C00005revised_csp_2_signed_31March%2016_REDACTED.PDF
- See also: D5160C00005_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1901&filename=D5160C00005_CSR_Synopsis_pdf..pdf